CLINICAL TRIAL: NCT01207362
Title: Assessing and Improving Balance Using Platform Perturbations
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Kevin Terry, PI, Kessler Foundation Research Center
Other Study IDs: R-648-09
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-09

CONDITIONS: Balance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Young adult
- Older adult

SUMMARY:
The purpose of this study is to compare current standing balance assessment methods to a new method that measures weight shift during small movements of a sliding platform. It will also be used to determine if balance improves with repeated exposure as part of a 4-week training program.

ELIGIBILITY:
Inclusion Criteria:

* Healthy no balance deficits age 20-35 or 50-65

Exclusion Criteria:

* moderate to severe arthritis

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-08 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in static sway | 20 days

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation Research Center, West Orange, New Jersey, United States